CLINICAL TRIAL: NCT01251848
Title: A Phase 1, Open Label, Randomized, Multiple Dose Study To Assess The Two-Way Drug Interaction Between Sitaxsentan And Low Dose Ritonavir In Healthy Subjects
Brief Title: Drug Interaction Between Ritonavir And Sitaxsentan
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1321061
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Sitaxentan; ritonavir; drug interaction; pharmacokinetics
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — sitaxsentan; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Active Comparator)
  Interventions: Drug: Sitaxentan
- Treatment B (Active Comparator)
  Interventions: Drug: Ritonavir
- Treatment C (Experimental)
  Interventions: Drug: Sitaxsentan; Drug: Ritonavir

INTERVENTIONS:
Drug: Sitaxentan — Sitaxsentan Tablet, 100 mg, q24h (once daily) for 5 days.
  Arms: Treatment A
Drug: Ritonavir — Ritonavir Capsule, 100 mg, q12h (twice daily) for 5 days (morning dose only on Day 5).
  Arms: Treatment B
Drug: Sitaxsentan — Sitaxsentan Tablet, 100 mg, q24h (once daily) for 5 days
  Arms: Treatment C
Drug: Ritonavir — Ritonavir Capsule, 100 mg, q12h (twice daily) for 5 days
  Arms: Treatment C

SUMMARY:
The study is to assess if sitaxsentan and ritonavir will affect the blood levels of each other when coadministered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or women of non-child bearing potential.
* Subjects (because of teratogenic risk of sitaxsentan) between the ages of 21 and 55 years, inclusive.
* Signed informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History of significant alcohol and drug use.
* Has hepatic dysfunction.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
The comparison of peak plasma concentration of sitaxsentan when coadministered with ritonavir versus sitaxsentan administered alone. | 24 hours
The comparison of area under the curve of sitaxsentan when coadministered with ritonavir versus sitaxsentan administered alone. | 24 hours
The comparison of peak plasma concentration of ritonavir when coadministered with sitaxsentan versus ritonavir administered alone. | 24 hours
The comparison of area under the curve of ritonavir when coadministered with sitaxsentan versus ritonavir administered alone. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321061&StudyName=Drug%20Interaction%20Between%20Ritonavir%20And%20Sitaxsentan%20